CLINICAL TRIAL: NCT00415441
Title: Efficacy and Cost-effectiveness of Physiotherapy for Chronic Rotator Cuff Pathology
Brief Title: Effectiveness of Physiotherapy for Chronic Shoulder Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Principal Investigator, Kim Bennell, Professor, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 299890
Record Dates: First submitted 2006-12-21; First posted 2006-12-22 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Shoulder Pain
Keywords: physiotherapy; exercise; manual therapy; shoulder pain; rotator cuff
MeSH Terms: conditions — Shoulder Pain; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active physiotherapy (Experimental): Manual therapy and home exercise program
  Interventions: Procedure: Physiotherapy program
- Placebo physiotherapy (Placebo Comparator): Manual therapy and home exercise program
  Interventions: Procedure: Placebo physiotherapy treatment

INTERVENTIONS:
Procedure: Physiotherapy program
  Arms: Active physiotherapy
Procedure: Placebo physiotherapy treatment
  Arms: Placebo physiotherapy

SUMMARY:
The purpose of this study is to investigate whether a physiotherapy program reduces pain and improves disability and quality-of-life in people with chronic shoulder pain.

The main study hypotheses are that (i) A 10-week physiotherapy treatment will result in significantly greater reductions in pain and disability than placebo treatment in individuals with chronic shoulder pain (ii) Improvements in pain and disability following a 10-week physiotherapy treatment will be maintained at a 3-month follow-up.

DETAILED DESCRIPTION:
Chronic rotator cuff pathology (CRCP) is a common cause of musculoskeletal morbidity in the community. Physiotherapy is often the first line of management for this condition. However, the effectiveness of physiotherapy for CRCP has not been well studied. Thus this project primarily aims to investigate the effect of a multimodality physiotherapy program to treat CRCP where effect is measured in terms of pain, disability and health-related quality of life. The secondary aim is to evaluate the cost-effectiveness of physiotherapy as a treatment for CRCP.

Comparison: physiotherapy program comprising stretches, exercises, manual techniques versus placebo physiotherapy

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of CRCP as evident by symptoms and signs including pain on active abduction or external rotation and positive impingement test;
* symptoms of pain in shoulder for > 3 months;
* average movement pain > 3 on a 10 cm visual analogue scale;
* aged ≥ 18 years;
* able to understand written and spoken English.

Exclusion Criteria:

* severe pain at rest, defined as > 7 on a visual analogue scale;
* global restriction of shoulder movements;
* systemic inflammatory joint disease;
* x-ray evidence of shoulder osteoarthritis or fracture;
* calcification about the shoulder joint;
* reason to suspect a complete rotator cuff rupture (eg. weakness of arm elevation, a positive "drop arm sign", a high riding humerus visible on x-ray or a complete tear on ultrasound);
* previous shoulder surgery on affected arm;
* physiotherapy, corticosteroid injection or hydrodilatation for shoulder in past 3 months;
* commenced non-steroidal antiinflammatory medication (NSAIDs) or conservative intervention in past 2 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2004-03; Primary Completion 2008-06 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index | Baseline and 11 weeks
Participant perceived global rating of change post treatment | 11 weeks

SECONDARY OUTCOMES:
Shoulder Pain and Disability Index at followup | 22 weeks
Participant perceived global rating of change at followup | 22 weeks
Australian Quality of Life Index at followup | Baseline, 11 weeks and 22 weeks
Isometric Shoulder strength using manual muscle tester post treatment and followup | Baseline, 11 weeks and 22 weeks
Participant assessment of average pain and restriction of activity post treatment and followup | Baseline, 11 weeks and 22 weeks
Cost effectiveness analysis | Baseline, 11 weeks and 22 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kim L Bennell, PhD, Principal Investigator — University of Melbourne, Australia; Rachelle Buchbinder, MPH, Principal Investigator — Monash University, Australia; Sally Green, PhD, Principal Investigator — Monash University; Anthony Harris, Principal Investigator — Monash University; Andrew Forbes, Principal Investigator — Monash University
Locations (1):
- University of Melbourne, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Bennell K, Wee E, Coburn S, Green S, Harris A, Staples M, Forbes A, Buchbinder R. Efficacy of standardised manual therapy and home exercise programme for chronic rotator cuff disease: randomised placebo controlled trial. BMJ. 2010 Jun 8;340:c2756. doi: 10.1136/bmj.c2756. PMID 20530557
- [Derived] Bennell K, Coburn S, Wee E, Green S, Harris A, Forbes A, Buchbinder R. Efficacy and cost-effectiveness of a physiotherapy program for chronic rotator cuff pathology: a protocol for a randomised, double-blind, placebo-controlled trial. BMC Musculoskelet Disord. 2007 Aug 31;8:86. doi: 10.1186/1471-2474-8-86. PMID 17761004